CLINICAL TRIAL: NCT00787735
Title: Services Research: Psychiatric Comorbidity in Drug Abuse
Brief Title: Improving Delivery of Mental Health Services for Patients With Drug Use and Other Behavioral and Emotional Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Robert Brooner, Professor of Psychiatry and Behavioral Sciences, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA016375 (NIH); R01DA016375 (NIH)
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Study Focusing on Integrated Versus Non-integrated Psychiatric Care in; Opioid-dependent and Methadone Treated Patients With Other Psychiatric; Diagnoses
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated Care (Experimental): Integrated Substance Abuse and Psychiatric Care (ISAP). Subjects received both their substance abuse and psychiatric care within the ATS clinic. Counseling compliance will be measured over time.
  Interventions: Behavioral: Counseling compliance
- Parallel Care (Active Comparator): Parallel Substance Abuse and Psychiatric Care (PSAP). Subjects received their substance abuse treatment at the ATS clinic. Their psychiatric care was received at Community Psychiatry. Counseling compliance will be measured over time.
  Interventions: Behavioral: Counseling compliance

INTERVENTIONS:
Behavioral: Counseling compliance — Rates of attendance to call counseling session over specific time points

SUMMARY:
This research is being done to:

* identify any emotional, behavioral or other troubling psychological problems that some people have who are seeking and receiving treatment for heroin or other drug use problems,
* learn if providing additional psychiatric treatment services in the ATS drug abuse treatment program is as beneficial for and acceptable to patients as referring them to the Bayview Community Psychiatry Program to get help for their emotional, behavioral and other psychological problems.

DETAILED DESCRIPTION:
This study will rigorously and systematically evaluate an integrated service delivery approach using a design that reduces many of the methodological limitations in earlier work. Study participants will include opioid abusers with a current psychiatric disorder. All study participants will receive comprehensive drug abuse treatment that includes adequate daily doses of methadone. Study participants will be randomly assigned to either an onsite and fully Integrated Substance Abuse and Psychiatric Care condition (ISAP-Integrated) or an offsite and non-integrated Parallel Substance Abuse and Psychiatric Care condition (PSAP-Parallel). Patients assigned to the ISAP condition will receive all of their ambulatory psychiatric care in the ATS treatment program; those assigned to the PSAP condition will be referred for matched "doses" of psychiatric care to the Community Psychiatry Program, which is located on the same campus as the ATS program. All drug abuse treatment services will be provided in the ATS program. Patients will be evaluated for 12 months on a range of outcome measures, including psychiatric medication and therapy adherence, drug abuse treatment adherence, changes in psychiatric symptoms, including posttraumatic stress disorder (PTSD), drug use, exposure to traumatic events, psychosocial functioning, and retention in both psychiatric and drug abuse treatment.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for current opioid physical dependence
* SAMSA Center for Substance Abuse Treatment - CSAT guidelines for maintenance on methadone or another approved opioid agonist
* have a current DSM-IV psychiatric disorder that is eligible for reimbursement in the Health Choice, Public Mental Health System (e.g., schizophrenia, mood disorders, anxiety disorders, personality disorders, adjustment disorder)
* express an interest in receiving psychiatric treatment for the problem.

Exclusion Criteria:

* pregnant
* acute medical problem that requires immediate and intense management (e.g., AIDS defining illness, tuberculosis, other serious and unstable medical disorder)
* delirium, dementia or mental retardation
* already receiving standard outpatient psychiatric care

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2004-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Days to first psychiatric appointment | within first 90 days of randomized care
Overall psychiatric counseling attendance compliance rate | 90, 180, and up to 365 days
  Includes attendance to all of the following sessions: psychiatrist, individual psychiatric counseling, and group psychiatric counseling.
Psychiatrist session attendance compliance rate | 90, 180, and up to 365 days
Individual and group psychiatric session attendance compliance rate | 90, 180, and up to 365 days

SECONDARY OUTCOMES:
Level of psychiatric distress | 90, 180, and up to 365 days
  Measured monthly using the Symptom Checklist 90-Revised (SCL90)
Urinalysis results | 90, 180, and up to 365 days
  Urinalysis tests are collected weekly. Results include tests for opioids, cocaine, benzodiazepines, and cannabis.

CONTACTS AND LOCATIONS:
Overall Officials: Robert K Brooner, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Addiction Treatment Services, Baltimore, Maryland, United States

REFERENCES:
- [Derived] King VL, Brooner RK, Peirce J, Kolodner K, Kidorf M. Challenges and outcomes of parallel care for patients with co-occurring psychiatric disorder in methadone maintenance treatment. J Dual Diagn. 2014;10(2):60-7. doi: 10.1080/15504263.2014.906132. PMID 24976801